CLINICAL TRIAL: NCT01258036
Title: Rôle de la Microarchitecture Osseuse Dans le déterminisme héréditaire de la fragilité Osseuse
Brief Title: Mother Daughter Bone Microarchitecture
Acronym: MODAM
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C09-37; 2009-A01295-52 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-03-18; First posted 2010-12-10 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Bone Fragility
Keywords: Bone microarchitecture; Bone mineral density; Bone markers; hereditary determinism
MeSH Terms: interventions — Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum plasma urine whole blood for DNA extraction
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fractured Mothers: Fractured Mothers and their daughters
  Interventions: Radiation: HRpQCT; Biological: Sampling; Radiation: Bone absorptiometry
- Non fractured mothers: Mothers non fractured and their daughters
  Interventions: Radiation: HRpQCT; Biological: Sampling; Radiation: Bone absorptiometry

INTERVENTIONS:
Radiation: HRpQCT — High Resolution peripheral Quantitative Computerized tomography
  Other Names: XTreme CT,Scanco Medical, Bassersdorf, Switzerland
Biological: Sampling — Urine and blood samples
  Other Names: Bone markers, hormones
Radiation: Bone absorptiometry — DXA at the lumbar spine, hip, radius and whole body
  Other Names: Hologic, Waltham,MA, USA

SUMMARY:
The aim of this study is to analyze the hereditary determinism of bone microarchitecture measured at the distal radius and distal tibia from a case control-study of mother-daughter pairs.

DETAILED DESCRIPTION:
Many factors influence the risk of osteoporosis but one of the most important is a positive family history, emphasizing the importance of genetics in the pathogenesis of osteoporosis. Till now, most genetic studies in osteoporosis have focused on the phenotype of BMD. However, areal BMD (bone quantity per unit bone area measured) does not provide information regarding bone distribution (between cortical and cancellous compartments) or bone microarchitecture (trabecular number, thickness, spacing and distribution) and cortical (thickness, porosity). We are planning to analyze the hereditary determinism of bone microarchitecture assessed non invasively with HR pQCT at the distal radius and the distal tibia in a case-control study with fractured and not fractured mothers and their daughters. Additionally, the role of the bone turnover, hormones involved in regulating bone metabolism , bone geometry measured at the proximal femur and bone strength estimated by finite element analysis (μFE)in the hereditary determinism of bone fragility will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Case mothers: postmenopausal women who have at least one bone fragility fracture confirmed by radiological examination or by a surgical report. Fragility fracture is a fracture that occurs as a result of a fall from standing height or less. Fractures of the skull, fingers and toes will be excluded.
* Control mothers: menopausal women not having suffered from bone fragility fracture.
* Daughters: Women aged 20 and older (postmenopausal or not), biological daughters of participating mothers. Several daughters from the same mother may be included.

Mothers and some daughters are recruited from the OFELY (Os des FEmmes de LYon) cohort or the FMC (Filière MédicoChirurgicale).

Exclusion Criteria:

* Adoptive daughters
* Nonmenopausal mothers

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Fractured mothers and their daughters (case group)
  2. Non-fractured mothers and their daughters (control group)
Sampling Method: Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

PRIMARY OUTCOMES:
Role of bone microarchitecture in the hereditary determinism of bone fragility | 18 months
  Comparison of bone microarchitecture parameters from high resolution peripheral quantitative computer tomography (HRpQCT)between daughters according to the fracture status of their mother.

SECONDARY OUTCOMES:
Role of Bone mineral density in the hereditary determinism of bone fragility | 18 months
  Comparison of BMD from DXA at the hip, the lumbar spine, the forearm and whole body, between daughters according to the fracture status of their mother.
Role of bone turnover and hormones in the hereditary determinism of bone fragility | 24 months
  Comparison of Bone markers and hormone levels between daughters according to the fracture status of their mother.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Sornay-Rendu, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Roland D Chapurlat, MD PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Unité Inserm 831, Pavillon F, Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Nagy H, Sornay-Rendu E, Boutroy S, Vilayphiou N, Szulc P, Chapurlat R. Impaired trabecular and cortical microarchitecture in daughters of women with osteoporotic fracture: the MODAM study. Osteoporos Int. 2013 Jun;24(6):1881-9. doi: 10.1007/s00198-012-2223-3. Epub 2012 Nov 23. PMID 23179577